CLINICAL TRIAL: NCT01056614
Title: Conditioning for Hematopoietic Cell Transplantation With Fludarabine Plus Targeted IV Busulfan and GVHD Prophylaxis With Thymoglobulin, Tacrolimus and Methotrexate in Patients With Myeloid Malignancies
Brief Title: Fludarabine Phosphate, Busulfan, and Anti-Thymocyte Globulin Followed By Donor Peripheral Blood Stem Cell Transplant, Tacrolimus, and Methotrexate in Treating Patients With Myeloid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1913.00; NCI-2009-01785 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1913.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P01HL036444 (NIH)
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Blastic Phase Chronic Myelogenous Leukemia; Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Myelodysplastic Syndromes; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Hematopoietic/Lymphoid Cancer; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Hematologic Neoplasms; Myeloproliferative Disorders; Leukemia, Myeloid, Acute | interventions — fludarabine phosphate; Busulfan; Antilymphocyte Serum; thymoglobulin; Tacrolimus; Methotrexate; merphos; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, PBSC transplant) (Experimental): Patients receive fludarabine phosphate IV over 30 minutes on days -9 to -6, busulfan IV over 3 hours on days -5 to -2, and anti-thymocyte globulin IV over 6 hours on days -3 and -2 and over 4 hours on day -1. Patients undergo allogeneic PBSC transplant on day 0. Patients then receive tacrolimus IV continuously or PO every 12 hours beginning on day -1 and taper to day 180 and methotrexate IV on days 1, 3, 6, and 11.
  Interventions: Drug: fludarabine phosphate; Drug: busulfan; Biological: anti-thymocyte globulin; Drug: tacrolimus; Drug: methotrexate; Procedure: peripheral blood stem cell transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: busulfan — Given IV
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
Biological: anti-thymocyte globulin — Given IV
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin
Drug: tacrolimus — Given IV and orally
  Other Names: FK 506; Prograf
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic PBSC transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic PBSC transplant
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying the side effects and how well giving fludarabine phosphate, busulfan, anti-thymocyte globulin followed by donor peripheral blood stem cell transplant, tacrolimus, and methotrexate works in treating patients with myeloid malignancies. Giving chemotherapy, such as fludarabine phosphate and busulfan, before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving anti-thymocyte globulin before transplant and tacrolimus and methotrexate after transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the incidence and severity of acute graft-versus-host disease (GvHD).

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics of intravenous (IV) busulfan including interdose variability and evaluation of a limited sampling strategy.

II. Determine thymoglobulin (anti-thymocyte globulin) pharmacokinetics.

III. Determine the incidence of donor engraftment.

IV. Determine system toxicities >= grade 3 per Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 3.

V. Determine the incidence and severity of chronic GvHD.

VI. Determine the incidence of non-relapse mortality at day +100 and at 1 year (yr).

VII. Determine the incidence of relapse.

VIII. Determine relapse-free survival.

IX. Determine the incidence of Epstein-Barr virus (EBV) activation.

OUTLINE:

Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -9 to -6, busulfan IV over 3 hours on days -5 to -2, and anti-thymocyte globulin IV over 6 hours on days -3 and -2 and over 4 hours on day -1. Patients undergo allogeneic peripheral blood stem cell (PBSC) transplant on day 0. Patients then receive tacrolimus IV continuously or orally (PO) every 12 hours beginning on day -1 and taper to day 180 and methotrexate IV on days 1, 3, 6, and 11.

After completion of study treatment, patients are followed at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Chronic myelogenous leukemia in chronic phase, accelerated phase and treated blast phase (CP2)
* Acute myeloid leukemia (AML) in remission or early relapse (< 10% marrow blasts)
* Myelodysplastic syndromes (MDS) ( all risk groups)
* Other myeloproliferative disorders
* DONOR: related or unrelated donors matched for human leukocyte antigen (HLA)-A, B, C, DRB1, and DQB1 defined by high resolution deoxyribonucleic acid (DNA) typing or mismatched for a single HLA-A, B, C, DRB1 or DQB1 allele
* DONOR: donor must consent to peripheral blood stem cell (PBSC) mobilization with granulocyte colony-stimulating factor (G-CSF) and leukapheresis; related donors will be collected at Fred Hutchinson Cancer Research Center (FHCRC), while unrelated donors will be collected through the National Marrow Donor Program (NMDP) or other donor centers
* DONOR: Age 12-75 yrs

Exclusion Criteria:

* Cardiac insufficiency requiring treatment or symptomatic coronary artery disease
* Hepatic disease, with aspartate aminotransferase (AST) > 2 times normal
* Severe hypoxemia, oxygen partial pressure (pO2) < 70 mm Hg, with decreased diffusion capacity of carbon monoxide (DLCO) < 70% of predicted; or mild hypoxemia, pO2 < 80 mm Hg with severely decreased DLCO < 60% of predicted
* Impaired renal function (creatinine > 2 times normal or estimated creatinine clearance < 60 ml/min)

  * MALE: ([140 -age in years] x ideal body weight [kg])/72 x serum creatinine (SCr) (mg/dL)
  * FEMALE: .85 x ([140-age in years] x ideal body weight [kg])/72 x SCr (mg/dL)
* Human immunodeficiency virus (HIV)-positive patients due to risk of reactivation or acceleration of HIV replication
* Female patients who are pregnant or breast feeding
* Life expectancy severely limited by diseases other than malignancy
* DONOR: donors who for any reason are unable to tolerate the mobilization and leukapheresis procedure
* DONOR: donors who are HIV-positive, or hepatitis B or C antigen-positive
* DONOR: female donors who have a positive pregnancy test

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2004-09; Primary Completion 2005-08 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Incidence of acute GvHD | Day 100 post-transplant
  Maximum grade of acute GVHD and the number of therapies required to treat GVHD will be determined.

SECONDARY OUTCOMES:
Pharmacokinetics of IV busulfan including interdose variability and evaluation of a limited sampling strategy | At 3.25, 4.5, 6, 8, 11, and 24-hours after the beginning of infusion on days -5, -4, and -3
Thymoglobulin pharmacokinetics | On day -3 prior to the first dose, on day -1 one hour after completion of infusion and on day 1 at 0900
Incidence of donor cell engraftment | By day 100
Incidence of system toxicities >= grade 3 as graded per CTCAE v.3 | Up to day 100 after transplantation
Incidence of chronic GvHD | Day 100
Incidence of non-relapse mortality defined as death without history of post-transplant relapse | At day 100
Incidence of non-relapse mortality defined as death without history of post-transplant relapse | At 1 year
Incidence of relapse | At 1 year
  Defined by either morphological or cytogenetic evidence of chronic myelogenous leukemia (CML), AML, MDS or other myeloproliferative disease in marrow, blood, or other sites, or laboratory evidence of residual disease.
Relapse-free survival | At 1 year
Incidence of EBV activation defined as an increase in plasma EBV DNA to >= 1000 copies/mL as determined by quantitative polymerase chain reaction (PCR) | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: H. Joachim Deeg, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States